CLINICAL TRIAL: NCT02042690
Title: Phase III Study to Compare Haplo-identical HSCT Versus Chemotherapy in First Remission for Standard-risk Adult Acute Lymphoblastic Leukemia
Brief Title: Haplo-identical HSCT Versus Chemotherapy for Adult Acute Lymphoblastic Leukemia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Chinese PLA General Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Peking University Aerospace Center Hospital (Other)
Responsible Party: Principal Investigator, Xiao-jun Huang,MD, Peking University People's Hospital, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALL-13
Record Dates: First submitted 2013-11-29; First posted 2014-01-23 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; hematopoietic stem cell transplantation; chemotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Drug Therapy; Methotrexate; Cyclophosphamide; Epirubicin; Dexamethasone; Mercaptopurine; Vindesine

STUDY DESIGN:
Intervention Model Description: After 1 year of enrollment, randomization was terminated because of the patients's intention to crossover between the two intervention groups (total enrolled n=16). The sample size was recalculated in July 2015, and the ethics committee agreed to modify the randomization scheme to intention-to-therapy (ITT). Patients who met the recruitment criteria after the second consolidation participated fully in discussions with their doctors and then made decisions on their own regarding their intention to receive haplo-SCT. For each patient, informed consent was obtained from that patient or his/her guardian in accordance with the Declaration of Helsinki.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chemotherapy (Active Comparator): Drugs:
  Drug:Methotrexate 1g/m2 d1,IV (in the vein) , used in cycle 1,3,5 Drug:arabinoside 2-3g/m2,q12h, d2-3, IV, used in cycle 1,3,5 Drug:cyclophosphamide:300mg/m2 q12h, d1-3, IV,used in cycle 2,4,6 Drug:Epirubicin 60mg/m2.d，d4,used in cycle 2,4,6 Drug:Vindesin 4mg/d，d4，d11, IV,in cycle 2,4,6 Drug:dexamethasone 40mg/d，d1-4，d11-14, IV, in cycle 2,4,6 Drug:Methotrexate 20 mg/m2/w,po, during maintenance treatment for 2 years Drug:6-mercaptopurine 60 mg/m2/d，po，d1-d28,during maintenance treatment for 2 years Drug:Vindesin 4mg/d，Predisone:1mg/kg, d1-7, every month during maintenance treatment for 2 years
  Interventions: Drug: Chemotherapy
- Haplo-identical HSCT (Experimental): Haplo-identical HSCT Protocol:G, donor treatment with recombinant granulocyte colony-stimulating factor (rhG-CSF); I, intensified immunologic suppression; A, antihuman thymocyte immunoglobulin (ATG) for the prevention of GVHD; C, combination of peripheral blood stem cell transplantation (PBSCT), and bone marrow transplantation (BMT)，named GIAC regimen. Graft versus-host disease(GVHD) prevention regimen: CSA/MMF/MTX, cyclosporine A(CSA) 1.25mg/kg/d, i.v administrated in two doses from day -109 until bowel function returned to normal, at which time patients receive oral CSA until 12months after HSCt and then gradually tapered. Every 12h, 0.5g mycophenolate mofetil (MMF)(0.25g for children) was administrated orally from day -10 to +30 and subsequently 0.25g from days +30 to +60. Methotrexate (MTX) was administrated at a dose of 15mg/m2 on day +1 and 10mg/m2 on days +3,+6, and +11.
  Interventions: Procedure: Haplo-identical HSCT

INTERVENTIONS:
Procedure: Haplo-identical HSCT — Haplo-identical Protocol: myeloablative human leukocyte antigen (HLA) haploidentical stem cell transplantation (haplo-SCT) using pretransplant ATG and granulocyte colony-stimulating factor (G-CSF)-stimulated grafts (ATG+G-CSF) GVHD prevention regimen: CSA/MMF/MTX, CSA 1.25mg/kg/d, i.v administrated in two doses from day -109 until bowel function returned to normal, at which time patients receive oral CSA until 12months after HRD-HSC and then gradually tapered. Every 12h, 0.5g MMF(0.25g for children) was administrated orally from day -10 to +30 and subsequently 0.25g from days +30 to +60. MTX was administrated at a dose of 15mg/m2 on day +1 and 10mg/m2 on days +3,+6, and +11.
  Arms: Haplo-identical HSCT
Drug: Chemotherapy — Patients receive 6 cycles of consolidation chemotherapy after randomization, including Hyper-CVAD-B regimen-Hyper-CVAD-A regimen/Hyper-CVAD-B regimen/Hyper-CVAD-A regimen/Hyper-CVAD-B regimen/Hyper-CVAD-A regimen.Maintenance treatment includes MTX 20mg/m2/w，po，6-mercaptopurine 60 mg/m2/d，po，d1-d28，VP（VDS 4mg,d1, Prednisone 1mg/kg d1-7) every one month for 2 years.
  Other Names: Methotrexate; arabinoside; cyclophosphamide; Epirubicin; dexamethasone; 6-mercaptopurine; Vindesin; Predisone
  Arms: chemotherapy

SUMMARY:
The survival of adult patients with standard-risk acute lymphoblastic leukemia(ALL) need to improve. We want to compare the efficacy of haplo-identical hematopoietic stem cell transplantation (HSCT) with chemotherapy for adult(age:18-39 years old) ALL patients in first phase of complete remission (CR1)

DETAILED DESCRIPTION:
Although the high complete remission rate (80%-90%) can be achieved, the long-term survival rate of standard-risk adult patients with acute lymphoblastic leukemia(ALL) is only 25%-55% when they receive chemotherapy alone. The survival rate can be further improved uo to 50%-75% when they receive HLA-matched HSCT However, the chance of finding a HLA-matched donor is low, especially in China. Alternative donor such as halpo-identical related donor might be an choice.

Our retrospective analysis showed about 59% overall survival could be achieved when standard-risk adult ALL patients received halpo-identical HSCT.Therefore, we start this randomization controlled trial to compare the efficacy of haplo-identical HSCT with chemotherapy for adult(age:18-39 years old) ALL patients in CR1.

ELIGIBILITY:
Inclusion Criteria:

* acute lymphoblastic leukemia
* 18-39 years old
* in first complete remission -Adequate hepatic function defined as: total bilirubin ≤2.0 times the institutional upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase(AST) ≤2.5 times the institutional ULN -
* Adequate renal function defined as creatinine ≤3 times the institutional ULN
* No uncontrollable infection
* Performance Status(PS)score 0-2(WHO)
* Subjects able to provide written informed consent

Exclusion Criteria:

* having HLA-matched donor
* high-risk ALL: (1)Ph+ALL (2)Hypodiploidy (3)t(v;11q23) (4) complex karyotype（≥5 chromosome abnormalities）（5）high white blood cell (WBC) count (B-ALL≥30×109/L;T-ALL ≥100×109/L).
* pregnancy
* Loss of ability to freely provide consent due to psychiatric or physical illness

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | At 2 years from study entry

SECONDARY OUTCOMES:
Rate of cumulative incidence of relapse | At 2 years from study entry
Overall survival (OS) rate | At 2 years from study entry
nonrelapse mortality | At 2 years from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peking University People's Hospital
Locations (5):
- China (5):
  - Aerospace Center Hospital, Beijing, Beijing Municipality
  - Wuhan Union Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - General Hospital of PLA, Beijing
  - Peking Union Hospital, Beijing

REFERENCES:
- [Derived] Lv M, Jiang Q, Zhou DB, Hu Y, Liu DH, Wu DP, Wang JB, Jiang H, Wang J, Chang YJ, Wang Y, Zhang XH, Xu LP, Liu KY, Huang XJ. Comparison of haplo-SCT and chemotherapy for young adults with standard-risk Ph-negative acute lymphoblastic leukemia in CR1. J Hematol Oncol. 2020 May 15;13(1):52. doi: 10.1186/s13045-020-00879-1. PMID 32414392